CLINICAL TRIAL: NCT06835322
Title: Effect of Finerenone on Proteinuria and GFR Progression in Patients With Non Diabetic Glomerulonephritis: A Randomized Clinical Trial
Brief Title: Effect of Finerenone in Patients With Non-diabetic Glomerulonephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Associate professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Finerenone and GN
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Glomerulonephritis
Keywords: finerenone; proteinuria; GFR progression; glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis; Proteinuria | interventions — finerenone

STUDY DESIGN:
Intervention Model Description: This research is a prospective randomized multicentric clinical trial in which 100 patients with biopsy proven glomerulonephritis (exception is nephrotic patients with positive anti-PLA2R indicative of primary membranous) will be randomly assigned to one of the study groups using block randomization with a ratio of 1:1.
  * Group A: 50 patients with biopsy proven glomerulonephritis who will receive 10 - 20 mg finerenone once daily orally in addition to their regular treatment protocol (RAAS blockers ± immunosuppression) for 6 months.
  * Group B: 50 patients with biopsy proven glomerulonephritis who will receive placebo once daily in addition to their regular treatment protocol (RAAS blockers ± immunosuppression) for 6 months.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): 50 patients with biopsy proven glomerulonephritis who will receive 10 - 20 mg finerenone once daily orally in addition to their regular treatment protocol (RAAS blockers ± immunosuppression) for 6 months.
  Interventions: Drug: Finerenone
- placebo (Placebo Comparator): 50 patients with biopsy proven glomerulonephritis who will receive placebo once daily in addition to their regular treatment protocol (RAAS blockers ± immunosuppression) for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone — 50 patients with biopsy proven glomerulonephritis who will receive 10 - 20 mg finerenone once daily orally in addition to their regular treatment protocol (RAAS blockers ± immunosuppression) for 6 months.
  Arms: interventional
Drug: Placebo — 50 patients with biopsy proven glomerulonephritis who will receive placebo once daily in addition to their regular treatment protocol (RAAS blockers ± immunosuppression) for 6 months.
  Arms: placebo

SUMMARY:
This study aims to assess the effect of finerenone on proteinuria and GFR progression in patients with non-diabetic glomerulonephritis.

DETAILED DESCRIPTION:
In patients with type 2 diabetes and advanced CKD, finerenone resulted in lower risks of CKD progression and cardiovascular events. Mineralocorticoid receptor over activation in the kidney leads to inflammation and fibrosis with subsequent progressive kidney disease. Finerenone, a nonsteroidal, selective mineralocorticoid receptor antagonist, had more potent anti-inflammatory and ant fibrotic effects than steroidal mineralocorticoid receptor antagonists. Finerenone has been shown to reduce the urinary albumin-to-creatinine ratio in patients with CKD treated with an RAS blocker, while having smaller effects on serum potassium levels than spironolactone.

Glomerulonephritis (GN) is an inflammation affecting kidney glomeruli, and is considered an important cause of CKD. Reducing proteinuria is one of the main therapeutic targets in patients with GN.

ELIGIBILITY:
Inclusion Criteria:

1. GN patients on maximum tolerated doses of an ACEi or ARBs together with their immunosuppression protocol (if needed) for at least 4 weeks.
2. urinary protein excretion >500 mg/g.
3. Adult patients with age above 18 years.
4. eGFR ≥ 25 mL/ min/1.73 m2.
5. baseline serum potassium level <5 mEq/L.

Exclusion Criteria:

1. Patients with diabetes mellitus (type 1 or 2).
2. Other non-glomerular kidney diseases.
3. Heart failure.
4. Breast feeding or pregnancy.
5. Patients who received medications to treat hyperkalemia 4 weeks before study.
6. Uncontrolled hypertension (BP > 160/100).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
- Change in kidney function | 6 months
  By assessing change in eGFR
- Change in proteinuria | 6 months
  By assessing change in protein to creatinine ratio
Change in kidney function | 6 months
  By assessing change in serum creatinine

SECONDARY OUTCOMES:
- Occurrence of hyperkalemia (potassium level >5 mEq/L) | 6 months
  By assessing serum K at baseline, then monthly
- Need for hospitalization | 6 months
  By assessing the need for hospital admission
- Serious adverse events | 6 months
  By reporting any serious adverse events during and after study for 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — Associate professor
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825
- [Background] Ruilope LM, Pitt B, Anker SD, Rossing P, Kovesdy CP, Pecoits-Filho R, Pergola P, Joseph A, Lage A, Mentenich N, Scheerer MF, Bakris GL. Kidney outcomes with finerenone: an analysis from the FIGARO-DKD study. Nephrol Dial Transplant. 2023 Feb 13;38(2):372-383. doi: 10.1093/ndt/gfac157. PMID 35451488
- [Background] Barrera-Chimal J, Girerd S, Jaisser F. Mineralocorticoid receptor antagonists and kidney diseases: pathophysiological basis. Kidney Int. 2019 Aug;96(2):302-319. doi: 10.1016/j.kint.2019.02.030. Epub 2019 Mar 13. PMID 31133455
- [Background] Grune J, Beyhoff N, Smeir E, Chudek R, Blumrich A, Ban Z, Brix S, Betz IR, Schupp M, Foryst-Ludwig A, Klopfleisch R, Stawowy P, Houtman R, Kolkhof P, Kintscher U. Selective Mineralocorticoid Receptor Cofactor Modulation as Molecular Basis for Finerenone's Antifibrotic Activity. Hypertension. 2018 Apr;71(4):599-608. doi: 10.1161/HYPERTENSIONAHA.117.10360. Epub 2018 Feb 5. PMID 29437893
- [Background] Bakris GL, Agarwal R, Chan JC, Cooper ME, Gansevoort RT, Haller H, Remuzzi G, Rossing P, Schmieder RE, Nowack C, Kolkhof P, Joseph A, Pieper A, Kimmeskamp-Kirschbaum N, Ruilope LM; Mineralocorticoid Receptor Antagonist Tolerability Study-Diabetic Nephropathy (ARTS-DN) Study Group. Effect of Finerenone on Albuminuria in Patients With Diabetic Nephropathy: A Randomized Clinical Trial. JAMA. 2015 Sep 1;314(9):884-94. doi: 10.1001/jama.2015.10081. PMID 26325557
- [Background] Hou JH, Zhu HX, Zhou ML, Le WB, Zeng CH, Liang SS, Xu F, Liang DD, Shao SJ, Liu Y, Liu ZH. Changes in the Spectrum of Kidney Diseases: An Analysis of 40,759 Biopsy-Proven Cases from 2003 to 2014 in China. Kidney Dis (Basel). 2018 Feb;4(1):10-19. doi: 10.1159/000484717. Epub 2017 Dec 8. PMID 29594138
- [Background] AlYousef A, AlSahow A, AlHelal B, Alqallaf A, Abdallah E, Abdellatif M, Nawar H, Elmahalawy R. Glomerulonephritis Histopathological Pattern Change. BMC Nephrol. 2020 May 18;21(1):186. doi: 10.1186/s12882-020-01836-3. PMID 32423387